CLINICAL TRIAL: NCT06939387
Title: Establishment, Evaluation and Treatment Strategy of Drug-induced Kidney Injury Model
Brief Title: Drug-induced Kidney Injury Model
Status: Recruiting | Type: Observational
Sponsor: Zhejiang Provincial People's Hospital (Other)
Collaborators: Taizhou Enze Medical Center Group (Other); Hangzhou Linping District first People's Hospital (Unknown); Aksu district first People's Hospital (Unknown); Ningbo Yinzhou District Second Hospital (Unknown); Wucheng District First People's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: KT2024116
Record Dates: First submitted 2025-03-10; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; drug
MeSH Terms: conditions — Acute Kidney Injury | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Drug induced acute kidney injury: Patients with acute kidney injury caused by the use of nephrotoxic drugs
  Interventions: Other: Observational study, no intervention

INTERVENTIONS:
Other: Observational study, no intervention — Observational study, no intervention

SUMMARY:
To establish the prediction model of renal dysfunction in patients with drug-induced renal injury and study the prognosis of different drug treatments

ELIGIBILITY:
Inclusion Criteria:

* Drug-induce acute kidney injury

Exclusion Criteria:

* 1.Dialysis patients; 2.No baseline creatinine; 3.Obstructive AKI; 4.Clinical data were incomplete.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Drug-induced acute kidney injury
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Model performance metrics assessed by AUC-ROC, accuracy and F1-score using 10-fold cross-validation | through study completion, an average of 6 months
  The prognosis of renal function was evaluated by measuring creatinine and proteinuria by laboratory tests. Predict outcomes using machine learning methods. And the prediction effect of the prediction model was evaluated by AUC-ROC, F1, accuracy and other indicators.

SECONDARY OUTCOMES:
The rate at which creatinine falls | 7 days, 1 month, 3 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
We will publish relevant research papers, patient data is not appropriate for public disclosure